CLINICAL TRIAL: NCT03355105
Title: Comparison of Two Methods of Adjusting the Mechanical In-Exsuflation in Neuromuscular Adult Patients
Acronym: EXSUFLOW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: K160910J; 2017-A01794-49 (Other: ANSM)
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Neuromuscular Diseases
Keywords: Neuromuscular disease
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Objective adjustment of the MI/E exsuflation pressure (Experimental): Objective adjustment of the MI/E exsuflation pressure based on the flow-volume curve generated during the cough.
  Interventions: Other: Objective adjustment of the MI/E exsuflation pressure and evaluation of cough effort
- Subjective adjustment of the MI/E exsuflation pressure (Active Comparator): Subjective adjustment of the MI/E exsuflation pressure based on the clinical judgment of the therapist and the patient.
  Interventions: Other: Subjective adjustment of the MI/E exsuflation pressure and evaluation of cough effort

INTERVENTIONS:
Other: Objective adjustment of the MI/E exsuflation pressure and evaluation of cough effort — The exsufflation pressures will be progressively increased starting from -20 cmH2O with 10 cmH2O increments up. 3 coughing operations will be realised for each level, until obtention of 10% of AUC decrease or a PCF collapse of at least 10% over the last 2 levels and without exceeding -70 cmH2O. The selected landing will be the one allowing the largest PCF without presence of collapse. An intermediate bearing between 2 bearings may be tested in order to approach an optimum adjustment threshold less than 5 cmH2O.
  Arms: Objective adjustment of the MI/E exsuflation pressure
Other: Subjective adjustment of the MI/E exsuflation pressure and evaluation of cough effort — The exsufflation pressures will be gradually increased from -20 cmH2O, with 10 cmH2O increments up to a maximum of -70 cmH2O. The selected level will be the one selected both by the patient and the "clinician" therapist and considered as making it possible to obtain the most effective cough according to the return of the patient.
  Arms: Subjective adjustment of the MI/E exsuflation pressure

SUMMARY:
In the context of neuromuscular diseases, the weakness of the respiratory muscles makes difficult to manage periods of congestion due to a less effective cough. It exposes the patient to bronchial superinfections that may require hospitalization. The use of cough assistance is therefore essential in order to avoid acute situations such as bronchial superinfections. Mechanical Insuflation-Exsufflation (MI / E) is an instrumental technique commonly used by therapists in a hospital or at the patient's home in order to facilitate the airway mucus clearance. The choice of the pressure settings of the IM / E is a decisive point because it conditions the effectiveness of the generated cough. It'is important to take into account the presence of any collapse in the use of IM / E in order to ensure the most effective cough given by the patient. Actually, except the common impression of the physiotherapist and the patient, there is no "simple" way for detecting and objectifying the threshold of collapse in the upper airways.

The aim of this study is to compare two modalities for the regulation of the level of the MI-E exsufflation, taking into account the presence of a collapse: a subjective "S" adjustment based on the clinical judgment of the therapist and the patient and an objective "O" adjustment based on the flow-volume curve generated during the cough.

DETAILED DESCRIPTION:
This is a bicentric, prospective crossover, randomized, open label trial. The study will focus on 50 adult patients with stable neuromuscular conditions, outside the congestion period requiring cough help.

Patients will be recruited from among the neuromuscular disease patients followed for their respiratory management in the home ventilation unit of the Raymond Poincaré Hospital Intensive care Unit or in the Aincourt Neurological Rehabilitation Service attached to the Vexin Intercommunal Hospital Group.

The cough help performed with the MI / E will be evaluated according to two conditions of adjustment of the exsufflation pressure: a subjective adjustment (modality S) and an objective adjustment (modality O), whose order will be randomized to control a phenomenon of tiredness causing confusion.

A respiratory technician and two therapists will participate to the protocol. The therapist "clinician" and "evaluator" role will be defined by a draw.

The protocol will take place during the same day of hospitalization in two stages:

* T0: validation of the eligibility criteria and inclusion of patients in the study.
* T1: evaluation of coughing performance according to the two modes of exsufflation pressure adjustment. Adjustment modality "S" according to the clinical impression of the "clinician" therapist and the patient, and the "Cough Peak Expiratory Flow" measured by the MI / E. Adjustment modality "O": according to the analysis of the flow / volume curve measured using a spirometer and a pneumotachograph.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Neuromuscular pathology
* Coughing aid information: DEPT <180 l / min
* In stable condition and without bulk
* Good understanding and cognition to follow the instructions and to inform the EVA
* Affiliated to a Sickness Insurance Plan or entitled
* Signed of informed consent

Exclusion Criteria:

* Pregnant woman
* Person under guardianship
* Inability to cooperate and / or communicate
* Acute decompensated organ
* Patient with following contraindications to mechanical in-exsufflation (MI-E) devices:

  1. pneumothorax
  2. pneumomediastinum
  3. pulmonary emphysema
  4. hemoptysis
  5. pleurisy
  6. nausea
  7. obstructive pulmonary disease or asthma
  8. recent lobectomy of the lung
  9. intracranial pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve (AUC) Flow Volume | At baseline
  The primary endpoint is the Area Under Curve (AUC) Flow Volume during the cough expiratory phase.
  To compare the cough effectiveness obtained according to the current modalities of the MI / E exsuflation pressure setting to that resulting from an adjustment based on the analysis of the flow-volume curve.

SECONDARY OUTCOMES:
Peak Cough Flow (PCF) | At baseline
  The Peak Cough Flow (PCF) : will be measured with a spirometer connected in series on the circuit of MI-E. Will be checked: whether the best AUC and the best PCF (regardless of the modality) occur during the same level of depression.
Evaluate the association between the peak cough flow (PCF) generated and the subjective criteria | At baseline
Subjective Therapist Cough Effectiveness | At baseline
  These measurements will be performed using an Analogical Visual Scale.
Subjective Patient Cough Effectiveness | At baseline
  These measurements will be performed using an Analogical Visual Scale.
Respiratory comfort | At baseline
  The respiratory comfort of the patient during the effort of cough. These measurements will be performed using an Analogical Visual Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric LOFASO, MD, PhD, Study Chair — Department of Physiology and Functional Explorations, Raymond Poincaré Hospital
Locations (1):
- Department of Physiology and Functional Explorations, Raymond Poincaré Hospital, Garches, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No